CLINICAL TRIAL: NCT01718704
Title: Study of Non-Invasive Viberect® Penile Vibratory Stimulation Regimen to Enhance Recovery of Erectile Function/Rigidity and Urinary Control/Continence After Nerve Sparing Radical Prostatectomy (RP) for Clinically Localized Prostate Cancer.
Brief Title: Viberect Penile Vibratory Stimulation to Enhance Recovery of Erectile Function and Urinary Continence Post-Prostatectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped due to inability to accrue patients because of competing trials.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00069795
Record Dates: First submitted 2012-10-24; First posted 2012-10-31 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Erectile Dysfunction Following Radical Prostatectomy; Urinary Incontinence of Non-organic Origin
Keywords: rehabilitation; erectile dysfunction; incontinence
MeSH Terms: conditions — Nocturnal Enuresis; Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Viberect device (Experimental): Men in this group will begin using the Viberect device 3 days after Foley catheter removal after surgery on a daily (or at least 4 times a week) basis for 7-10 minutes in a relaxed setting.
  Interventions: Device: Viberect device
- No Viberect (No Intervention): Men in this group will not be provided with the Viberect device

INTERVENTIONS:
Device: Viberect device — Men who begin using the Viberect device 3 days after Foley catheter removal on a daily (or at least 4 times a week) basis for 7-10 minutes in a relaxed setting with sexual thoughts or foreplay for one year. Viberect method can be performed by the person's sexual partner.
  Arms: Viberect device

SUMMARY:
The purpose of this study is to evaluate whether using penile vibratory stimulation with the Viberect handheld device can help the recovery of erections and urinary control after radical prostatectomy.

DETAILED DESCRIPTION:
Prostate cancer screening programs have led to thousands of sexually healthy and continent men being diagnosed with prostate cancer every year. Recent literature suggests that up to 80% of these cancers are confined to the prostate gland. Currently, radical prostatectomy (RP) remains the best option for management of clinically localized prostate cancer in men with life expectancy greater than 10 years. Despite providing optimal cancer control, surgery can lead to quality of life (QOL) problems such as urinary incontinence and erectile dysfunction (ED). Refinement of surgical technique have improved sexual and continence outcomes; however erectile function lags behind other QOL measures by 1-2 years, and quality of returning erections is often inferior. This can have profound biological, marital, and psychological consequences in potent men undergoing RP.

ED is the inability to develop and maintain an erection for satisfactory sexual intercourse or activity. ED after nerve-sparing RP is related to a certain degree with functional impairment of cavernous nerves (CN) that travel along the prostate to the penis. This neuropraxia can last as long as 2 years. Pro-erectile nerve stimulus is vital for replenishment of corporal oxygen supply and other metabolic needs. Several histological analyses have demonstrated decreased smooth muscle number, cell-cell contact, venous leakage, collagen deposition, and additional harmful effects to corporal tissue after injury to CN.

Awaiting post-surgical neuropraxia recovery, urologists have proposed a proactive approach to use of oral, intraurethral or injectable pharmacotherapy, neuromodulation, or vacuum-assisted regimens in erectile rehabilitation programs. Several studies demonstrate variable functional improvement in erectile function. Unfortunately, prohibitive costs of medications, poor response, and pain from injectables or intraurethral application often lead to high dropout rates.

In addition to ED, a significant proportion of men after surgery develop and suffer from urinary incontinence (Stress, Urge, Mixed) requiring wearing pads with bothersome complaints persisting for months, even years after RP.

The primary objective is to assess the role of penile vibratory stimulation by the Viberect device in enhancing the recovery of erectile function/rigidity and urinary continence after RP for clinically localized prostate cancer. The difference in penile length will be compared in each arm.

The secondary objective is to obtain a formal risk analysis (RA). Other objectives are to assess the ease of use and acceptability of vibratory stimulation at home.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven low/moderate risk prostate cancer (Gleason 3+3=6, 3+4=7, 3+2=5, 2+3=5, cT1c, cT2a, cT2b, preoperative prostatic specific antigen (PSA) less than 10)
* between ages 40-70
* preoperative IIEF (erectile function domain) score equal or greater than 20
* IPSS less than 10 and no urinary incontinence

Exclusion Criteria:

* Men with neurological disease
* IIEF score less than 20
* high risk prostate cancer (Gleason 4+3=7, 4+4=8, any Gleason 5, cT2c, cT3, PSA > 10)
* spinal cord injury
* history of transurethral resection of prostate (TURP) or other prostate ablative procedures
* history of priapism, pelvic neuropathy, penile skin lesions/ulcers
* inability to understand and demonstrate device use instructions.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
change in erectile function | baseline to 6 weeks after first device use
  The International Index for Erectile Function (IIEF) questionnaire will be administered. This is a 15 item tool; 6 ask questions addressing Erectile function over the previous 4 weeks. Scores from 0-30 can be obtained in this domain. Scores are interpreted as follows: 0-6 = Severe dysfunction, 7-12 = Moderate dysfunction, 13-18 = mild-moderate dysfunction, 19-24 = mild dysfunction, 25-30 = No dysfunction
change in erectile function | baseline to 3 months after first device use
  IIEF questionnaire will be administered. This is a 15 item tool; 6 ask questions addressing Erectile function over the previous 4 weeks. Scores from 0-30 can be obtained in this domain. Scores are interpreted as follows: 0-6 = Severe dysfunction, 7-12 = Moderate dysfunction, 13-18 = mild-moderate dysfunction, 19-24 = mild dysfunction, 25-30 = No dysfunction
change in erectile function | baseline to 6 months after first device use
  IIEF questionnaire will be administered. This is a 15 item tool; 6 ask questions addressing Erectile function over the previous 4 weeks. Scores from 0-30 can be obtained in this domain. Scores are interpreted as follows: 0-6 = Severe dysfunction, 7-12 = Moderate dysfunction, 13-18 = mild-moderate dysfunction, 19-24 = mild dysfunction, 25-30 = No dysfunction
change in erectile function | baseline to 9 months after first device use
  The International Index for Erectile Function (IIEF) questionnaire will be administered. This is a 15 item tool; 6 ask questions addressing Erectile function over the previous 4 weeks. Scores from 0-30 can be obtained in this domain. Scores are interpreted as follows: 0-6 = Severe dysfunction, 7-12 = Moderate dysfunction, 13-18 = mild-moderate dysfunction, 19-24 = mild dysfunction, 25-30 = No dysfunction
change in erectile function | baseline to 12 months after first device use
  The International Index for Erectile Function (IIEF) questionnaire will be administered. This is a 15 item tool; 6 ask questions addressing Erectile function over the previous 4 weeks. Scores from 0-30 can be obtained in this domain. Scores are interpreted as follows: 0-6 = Severe dysfunction, 7-12 = Moderate dysfunction, 13-18 = mild-moderate dysfunction, 19-24 = mild dysfunction, 25-30 = No dysfunction
change in erectile function | baseline to 6 weeks after first device use
  The Expanded Prostate Cancer Index Composite (EPIC) sexual assessment questionnaire will be administered. The tool has 9 questions about erectile function over the previous 4 weeks. It is scored from 9 - 43 with higher scores indicating greater dysfunction
change in erectile function | baseline to 3 months after first device use
  The Expanded Prostate Cancer Index Composite (EPIC) sexual assessment questionnaire will be administered. The tool has 9 questions about erectile function over the previous 4 weeks. It is scored from 9 - 43 with higher scores indicating greater dysfunction
change in erectile function | baseline to 6 months after first device use
  The Expanded Prostate Cancer Index Composite (EPIC) sexual assessment questionnaire will be administered. The tool has 9 questions about erectile function over the previous 4 weeks. It is scored from 9 - 43 with higher scores indicating greater dysfunction
change in erectile function | baseline to 9 months after first device use
  The Expanded Prostate Cancer Index Composite (EPIC) sexual assessment questionnaire will be administered. The tool has 9 questions about erectile function over the previous 4 weeks. It is scored from 9 - 43 with higher scores indicating greater dysfunction
change in erectile function | baseline to 12 months after first device use
  The Expanded Prostate Cancer Index Composite (EPIC) sexual assessment questionnaire will be administered. The tool has 9 questions about erectile function over the previous 4 weeks. It is scored from 9 - 43 with higher scores indicating greater dysfunction
change in erectile function | baseline to 6 weeks after first device use
  The Erectile Hardness Score (EHS) questionnaire will be administered. it is a single item tool. It is scored from 1 to 4. 4 indicates attainment of full rigidity with ability to perform penetrative intercourse
change in erectile function | baseline to 3 months after first device use
  The Erectile Hardness Score (EHS) questionnaire will be administered. it is a single item tool. It is scored from 1 to 4. 4 indicates attainment of full rigidity with ability to perform penetrative intercourse
change in erectile function | baseline to 6 months after first device use
  The Erectile Hardness Score (EHS) questionnaire will be administered. it is a single item tool. It is scored from 1 to 4. 4 indicates attainment of full rigidity with ability to perform penetrative intercourse
change in erectile function (EF) | baseline to 9 months after first device use
  The Erectile Hardness Score (EHS) questionnaire will be administered. it is a single item tool. It is scored from 1 to 4. 4 indicates attainment of full rigidity with ability to perform penetrative intercourse
change in EF | baseline to 12 months after first device use
  The Erectile Hardness Score (EHS) questionnaire will be administered. it is a single item tool. It is scored from 1 to 4. 4 indicates attainment of full rigidity with ability to perform penetrative intercourse
change in EF | baseline to 6 weeks after first device use
  Measurement of penile length from corona to dorsal glans penis in centimeters
change in EF | baseline to 3 months after first device use
  Measurement of penile length from corona to dorsal glans penis in centimeters
change in EF | baseline to 6 months after first device use
  Measurement of penile length from corona to dorsal glans penis in centimeters
change in EF | baseline to 9 months after first device use
  Measurement of penile length from corona to dorsal glans penis in centimeters
change in EF | baseline to 12 months after first device use
  Measurement of penile length from corona to dorsal glans penis in centimeters

SECONDARY OUTCOMES:
change in urinary control | baseline to 6 weeks after first device use
  The Expanded Prostate Cancer Index Composite (EPIC) urinary function assessment questionnaire will be administered. This is a 7 item tool assessing urinary function over the past 4 weeks. Higher scores indicate decreased urinary control
change in urinary control | baseline to 3 months after first device use
  The Expanded Prostate Cancer Index Composite (EPIC) urinary function assessment questionnaire will be administered. This is a 7 item tool assessing urinary function over the past 4 weeks. Higher scores indicate decreased urinary control
change in urinary control | baseline to 6 months after first device use
  The Expanded Prostate Cancer Index Composite (EPIC) urinary function assessment questionnaire will be administered. This is a 7 item tool assessing urinary function over the past 4 weeks. Higher scores indicate decreased urinary control
change in urinary control | baseline to 9 months after first device use
  The Expanded Prostate Cancer Index Composite (EPIC) urinary function assessment questionnaire will be administered. This is a 7 item tool assessing urinary function over the past 4 weeks. Higher scores indicate decreased urinary control
change in urinary control | baseline to 12 months after first device use
  The Expanded Prostate Cancer Index Composite (EPIC) urinary function assessment questionnaire will be administered. This is a 7 item tool assessing urinary function over the past 4 weeks. Higher scores indicate decreased urinary control
change in urinary control | baseline to 6 weeks after first device use
  Mass of incontinence guards used over a 24 hour period in grams
change in urinary control | baseline to 3 months after first device use
  Mass of incontinence guards used over a 24 hour period in grams
change in urinary control | baseline to 6 months after first device use
  Mass of incontinence guards used over a 24 hour period in grams
change in urinary control | baseline to 9 months after first device use
  Mass of incontinence guards used over a 24 hour period in grams
change in urinary control | baseline to 12 months after first device use
  Mass of incontinence guards used over a 24 hour period in grams
change in urinary control | baseline to 6 weeks after first device use
  The International Prostate Symptom Score (IPSS) Questionnaire will be administered. 7 questionnaires address urinary control with a total attainable score from 0-35. 0 = no dysfunction, 1-7 = mild dysfunction, 8 - 19 = moderate dysfunction, 20-35 = severe dysfunction. The 8th/final item addresses impact of urinary control on quality of life
change in urinary control | baseline to 3 months after first device use
  The International Prostate Symptom Score (IPSS) Questionnaire will be administered. 7 questionnaires address urinary control with a total attainable score from 0-35. 0 = no dysfunction, 1-7 = mild dysfunction, 8 - 19 = moderate dysfunction, 20-35 = severe dysfunction. The 8th/final item addresses impact of urinary control on quality of life
change in urinary control | baseline to 6 months after first device use
  The International Prostate Symptom Score (IPSS) Questionnaire will be administered. 7 questionnaires address urinary control with a total attainable score from 0-35. 0 = no dysfunction, 1-7 = mild dysfunction, 8 - 19 = moderate dysfunction, 20-35 = severe dysfunction. The 8th/final item addresses impact of urinary control on quality of life
change in urinary control | baseline to 9 months after first device use
  The International Prostate Symptom Score (IPSS) Questionnaire will be administered. 7 questionnaires address urinary control with a total attainable score from 0-35. 0 = no dysfunction, 1-7 = mild dysfunction, 8 - 19 = moderate dysfunction, 20-35 = severe dysfunction. The 8th/final item addresses impact of urinary control on quality of life
change in urinary control | baseline to 12 months after first device use
  The International Prostate Symptom Score (IPSS) Questionnaire will be administered. 7 questionnaires address urinary control with a total attainable score from 0-35. 0 = no dysfunction, 1-7 = mild dysfunction, 8 - 19 = moderate dysfunction, 20-35 = severe dysfunction. The 8th/final item addresses impact of urinary control on quality of life

OTHER OUTCOMES:
change in assessment of ease and acceptability of use of the Viberect | 6 weeks after first device use to 3 months
  The Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) questionnaire will be administered. This is an 11 item tool addressing participant satisfaction with the Viberect; higher scores indicate greater dissatisfaction
change in assessment of ease and acceptability of use of the Viberect | 6 weeks after first device use to 6 months
  The Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) questionnaire will be administered. This is an 11 item tool addressing participant satisfaction with the Viberect; higher scores indicate greater dissatisfaction
change in assessment of ease and acceptability of use of the Viberect | 6 weeks after first device use to 9 months
  The Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) questionnaire will be administered. This is an 11 item tool addressing participant satisfaction with the Viberect; higher scores indicate greater dissatisfaction
change in assessment of ease and acceptability of use of the Viberect | 6 weeks after first device use to 12 months
  The Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) questionnaire will be administered. This is an 11 item tool addressing participant satisfaction with the Viberect; higher scores indicate greater dissatisfaction
change in assessment of ease and acceptability of use of the Viberect | baseline to 6 weeks after first device use
  The Treatment Satisfaction Scale (TSS) questionnaire will be administered. This is an 21 item tool addressing participant satisfaction with the Viberect; higher scores indicate greater dissatisfaction
change in assessment of ease and acceptability of use of the Viberect | baseline to 3 months after first device use
  The Treatment Satisfaction Scale (TSS) questionnaire will be administered. This is an 21 item tool addressing participant satisfaction with the Viberect; higher scores indicate greater dissatisfaction
change in assessment of ease and acceptability of use of the Viberect | baseline to 6 months after first device use
  The Treatment Satisfaction Scale (TSS) questionnaire will be administered. This is an 21 item tool addressing participant satisfaction with the Viberect; higher scores indicate greater dissatisfaction
change in assessment of ease and acceptability of use of the Viberect | baseline to 9 months after first device use
  The Treatment Satisfaction Scale (TSS) questionnaire will be administered. This is an 21 item tool addressing participant satisfaction with the Viberect; higher scores indicate greater dissatisfaction
change in assessment of ease and acceptability of use of the Viberect | baseline to 12 months after first device use
  The Treatment Satisfaction Scale (TSS) questionnaire will be administered. This is an 21 item tool addressing participant satisfaction with the Viberect; higher scores indicate greater dissatisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Arthur L Burnett, MD, MBA, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Frederick Urology Specialists, Frederick, Maryland